CLINICAL TRIAL: NCT06225258
Title: Analysis of Anti-inflammatory Effect of Hop Extract Rich in Xanthohumol in Patients Treated for Septic Shock
Brief Title: Xanthohumol as an Adjuvant in the Treatment of Septic Shock
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEPXN
Record Dates: First submitted 2023-12-21; First posted 2024-01-25 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Septic Shock; Pneumonia; ARDS
Keywords: septic shock; inflammation; Xanthohumol; adjuvant; endotheliopathy; ARDS; cytokine
MeSH Terms: conditions — Shock, Septic; Pneumonia; Inflammation | interventions — xanthohumol

STUDY DESIGN:
Intervention Model Description: Patients are randomised in a double-blind, placebo-controlled manner to two groups using sealed envelopes. In the intervention group, all patients receive Xanthohumol as adjunctive therapy as recommended by the Surviving Sepsis Campaign. In the control group, patients are treated without Xanthohumol as recommended by the Surviving Sepsis Campaign and are treated as recommended by Surviving Sepsis.
  Bioavailability, clinical and possible side effects are monitored.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group C (No Intervention): Patients are treated according to the recommendations of the Surviving Sepsis Campaign.
- Group Xn (Experimental): Patients, who are admitted to the Intensive Care Unit (ICU) due to septic shock in the early, acute phase. Patients are treated according to the recommendations of the Surviving Sepsis Campaign and receive xanthohumol at a dose of 2 mg per kg body weight administered via nasogastric tube as supportive therapy.
  Interventions: Dietary Supplement: Xanthohumol

INTERVENTIONS:
Dietary Supplement: Xanthohumol — Patients, who received Xanthohumol (Chmiel-Xn-Active, SALUTIS Pharmacy, Poland) as adjunctive therapy to treatment recommended by Surviving Sepsis Campaign. Xanthohumol is administrated by the nosogastric tube three times a day *every 8 hours) at the dose of 2 mg.\/kg body weight for 10 days. The first dose of Xanthohumol is administrated within 4 hours after the admission to the ICU.
  Other Names: ChmielXnActive (Salutis Pharmacy, Poland)
  Arms: Group Xn

SUMMARY:
Septic shock (SS) is a life-threatening condition resulting from excessive inflammatory response to bacterial, viral or/and fungal infections. It is associated with dysregulation of the immune system, activation of immune cells, and massive release of cytokines, commonly known as the cytokine storm (CS). The clinical manifestations of SS depend on the initial site of infection. However, the classic symptoms are associated with severe dysfunction of the respiratory and cardiovascular systems, which are observed from the early phase. Respiratory insufficiency frequently requires different forms of oxygen supplementation, including mechanical ventilation and even extracorporeal oxygenation. The severity of respiratory and other organ dysfunction depends on the inflammatory response to the infection and circulating toxins, which correspond to excessive cytokine release. In the past years, several studies documented that reduction of SS-related inflammatory response and CS improved organ function and alleviated the clinical course of SS. Unfortunately, an effective strong anti-inflammatory without side effects medications has not yet been found. Therefore, the use of natural anti-inflammatory and antioxidant substances seems very promising.

Xanthohumol (Xn) is a natural prenylated chalcone extracted from the female inflorescences of hop cones (Humulus lupus) and possesses strong anti-inflammatory and antioxidant properties. It is widely used as a supplement to diet. Xanthohumol inhibits CS and has been showed to be an effective medication for reducing the severity of lung injury. It has been documented that Xn inhibits proinflammatory pathways in a different manner. A decrease in cytokine production and release can affect endothelial function and correct inflammatory-related vascular hyperpermeability, reducing uncontrolled water shift to extravascular space and then tissue edema. Clinical observation showed that administration of Xn alleviated clinical course, improved respiratory function, and reduced mortality in critically ill COVID-19 patients. Xanthohumol is safe and well tolerated by humans, and no adverse effects have been reported yet. Based on its strong anti-inflammatory and antioxidative properties, it can be speculated that the use of Xn can effectively reduce the inflammatory response and improve the clinical course in SS patients.

ELIGIBILITY:
Inclusion Criteria:

* a septic shock in the early, acute phase,
* respiratory insufficiency required mechanical ventilation with PaO2/FiO2 < 150,
* bacterial infection,
* procalcitonin higher than 5 ng/mL and interleukin 6 higher than 100 pg/mL,
* no allergy to hops or their derivatives,
* hemodynamic instability requiring vasopressor infusions

Exclusion Criteria:

* lack of agreement
* septic shock treated for more than 1 day,
* history of severe chronic cardiac, pulmonary and/or liver diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Xanthohumol as an adjunctive treatment improves clinical course in ill septic shock patents | 7 and 28 days mortality
  Xanthohumol as an adjunctive treatment can significantly reduce mortality and length of hospitalization in critically ill patients. This effect can be reflected by analysis of the mortality rate on days 7 and 28 after the admission to the ICU.
Xanthohumol as an adjunctive treatmenty affects a severity of inflammation | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  The use of xanthohumol as adjunctive treatment can reduce the inflammatory response in the acute early phase of septic shock. Plasma concentrations of pro-inflammatory cytokines can reflect this effect. Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.
Xanthohumol as an adjunctive treatment affects sepsis-related glycocalyx injury | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  The use of xanthohumol as adjunctive treatment can reduce septic-induced glycocalyx injury. The severity of glycocalyx damage can be measured by changes in plasma biomarker concentrations, which are typical of glycocalyx damage. Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.

SECONDARY OUTCOMES:
Xanthohumol as an adjunctive treatment affects plasma interleukin 1beta concentration. | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  Interleukin 1beta, also known as lymphocyte activating factor, is produced and released by activated macrophages and monocytes and is important biomarker of inflammatory response. Its elevated concentrations relate to severity of inflammation, while its reduction corresponds to effective treatment. Rapid decrease in the circulating interleukin 1beta concentration may confirm the efficacy of Xanthohumol in critically ill patients treated for septic shock.
  Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.
Xanthohumol as an adjunctive treatment changes plasma tumor necrosis factor-alpha concentration. | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  Tumor necrosis factor-alpha (TNF-alpha) is a pro-inflammatory cytokine released by different cells including macrophages, endothelial cells, lymphoid cells and others to stimulate the immune system into an inflammatory response. It is released as a response to lipopolysaccharide or other bacterial products following infection. A high concentration of TNF-alpha corresponds to the severity of inflammatory response and endothelial hyper-permeability with glycocalyx damage. Rapid decrease in the circulating TNF-alpha concentration may confirm the efficacy of Xanthohumol in critically ill patients treated for septic shock. Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.
Xanthohumol as an adjunctive treatment affects plasma interleukin 6 concentration. | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  Interleukin 6 is the most recognized pro-inflammatory cytokine. It is also anty-inflammatory myokine. Interleukine 6 is released by macrophages in response to microbial molecules such as pathogen-associated molecular patterns or damage-associated molecular patterns. Interleukin 6 is an important mediator of fever and of the acute phase of inflammatory response. A rapid decrease in the circulating interleukin 6 concentration may confirm the efficacy of Xanthohumol in critically ill patients treated for septic shock. Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.
Xanthohumol as an adjunctive treatment affects plasma interleukin 8 concentration. | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  Interleukin 8 is a chemokine produced by different cells including macrophages and epithelial cells. It is a mediator associated with inflammation and plays a crucial role in neutrophil recruitment and neutrophil degranulation. Interleukin 8 is secreted as a response to oxidant stress. It correlates with endothelial injury. Its rapid decrease in the circulating blood may confirm the efficacy of Xanthohumol in critically ill patients treated for septic shock. Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.
Xanthohumol as an adjunctive treatment affects plasma interleukin 17 concentration | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  Interleukin 17 is a pro-inflammatory cytokine that is produced by a group of T helper cells known as T helper 17 cells in response to their stimulation with interleukin 23. Its elevated concentrations correspond to the severity of inflammation, while its reduction corresponds to effective treatment. A decrease in its concentration in the circulating blood may confirm the efficacy of Xanthohumol in critically ill patients treated for septic shock. Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.
Xanthohumol as an adjunctive treatment affects plasma interleukin 23 concentration. | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  Interleukin 23 is an inflammatory cytokine secreted by activated dendric cells, macrophages, or monocytes. IL-23 is also produced by B cells through B cell antigen receptor signaling. Polarisation to a Th17 phenotype is triggered by interleukin-6. Rapid decrease in the circulating IL-23 concentration may reflect changes in IL-17 concentration that confirm the efficacy of Xanthohumol in critically ill patients treated for septic shock. Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.
Xanthohumol as an adjunctive treatment affects plasma interleukin 40 concentration | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  Interleukin 40 is synthetized by C17orf99 and activated B cells after being stimulated with anti-CD40 monoclonal antibodies. It is a key effector in the humoral immune system. IL-40 exerts proinflammatory effects. Decrease in IL-40 may confirm the efficacy of Xanthohumol in critically ill patients treated for septic shock. Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.
Xanthohumol as an adjunctive treatment affects plasma syndecan 1 concentration. | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  Syndecan-1 is a heparan sulfate proteoglycan expressed in endothelial cells and is a well-known marker of endothelial glycocalyx degradation. Its elevated plasma concentration corresponds to endothelial injury and was noted in septic shock patients. A decrease in the inflammatory response following Xanthohumol administration reduces the severity of glycocalyx damage and endothelial injury. Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.
Xanthohumol as an adjunctive treatment affects plasma vascular endothelial adhesion molecule 1 concentration. | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  Vascular endothelial adhesion molecule 1 is a protein expressed in endothelial cells in response to pro-inflammatory cytokines including interleukine1 and tumor necrosis factor-alpha or bacterial endotoxin. Its elevated plasma concentration correlates with disorders in vascular permeability and documents endothelial damage following inflammation. A decrease in the severity of inflammation and the amount of circulating pro-inflammatory cytokines can reduce the severity of endothelial injury reflected by a decrease in plasma vascular endothelial adhesion molecule 1 concentration. Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.
Xanthohumol as an adjunctive treatment affects plasma E-selectin concentration. | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  E-selectin is a glycoprotein expressed on endothelial cells after activation by interleukin 1beta, tumor necrosis factor-alpha, or bacterial lipopolysaccharides. Its expression is crucial to control leukocyte accumulation in inflammatory responses. Elevated plasma E-selectin concentration was documented in sepsis and patients treated for inflammatory diseases without septic syndromes. Plasma E-selectin concentration correlates with the severity of inflammation and endothelial damage. A decrease in the severity of inflammation and the amount of circulating pro-inflammatory cytokines can reduce the severity of endothelial injury reflected by a decrease in plasma vascular endothelial adhesion molecule 1 concentration. Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.
Xanthohumol as an adjunctive treatment affects plasma vascular endothelial growth factor concentration. | 7 time points: just after ICU admission and on the days 1,2,3,4,5 and 6 after ICU admission.
  Vascular endothelial growth factor (VEGF) is a protein, which is considered as a sensitive marker of endothelial damage and vascular permeability. It is originally known as vascular permeability factor. VEGF-A production can be induced in the endothelial cells by circulating cytokines and severe hypoxia. A decrease in the severity of inflammation and the amount of circulating pro-inflammatory cytokines can reduce the severity of endothelial injury reflected by a decrease in VEGF-A concentration. Blood samples are collected from arterial access at nine time points: just after ICU admission (baseline) and in the morning on days 1, 2, 3, 4, 5, and 6 after ICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Dabrowski, Prof, Study Chair — Medical University of Lublin, Poland; Wlodzimierz Plotek, Principal Investigator — Medical University of Lublin, Poland
Locations (1):
- Intensive Care Unit, University Hospital No 4,, Lublin, Lublin Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartmanska A, Tronina T, Poplonski J, Huszcza E. Biotransformations of prenylated hop flavonoids for drug discovery and production. Curr Drug Metab. 2013 Dec;14(10):1083-97. doi: 10.2174/1389200214666131211151855. PMID 24329115
- [Background] Bosmann M, Ward PA. The inflammatory response in sepsis. Trends Immunol. 2013 Mar;34(3):129-36. doi: 10.1016/j.it.2012.09.004. Epub 2012 Oct 2. PMID 23036432
- [Background] Chen X, Li Z, Hong H, Wang N, Chen J, Lu S, Zhang H, Zhang X, Bei C. Xanthohumol suppresses inflammation in chondrocytes and ameliorates osteoarthritis in mice. Biomed Pharmacother. 2021 May;137:111238. doi: 10.1016/j.biopha.2021.111238. Epub 2021 Jan 28. PMID 33517187
- [Background] Corrado C, Barreca MM, Raimondo S, Diana P, Pepe G, Basilicata MG, Conigliaro A, Alessandro R. Nobiletin and xanthohumol counteract the TNFalpha-mediated activation of endothelial cells through the inhibition of the NF-kappaB signaling pathway. Cell Biol Int. 2023 Mar;47(3):634-647. doi: 10.1002/cbin.11963. Epub 2022 Nov 15. PMID 36378586
- [Background] Costa R, Negrao R, Valente I, Castela A, Duarte D, Guardao L, Magalhaes PJ, Rodrigues JA, Guimaraes JT, Gomes P, Soares R. Xanthohumol modulates inflammation, oxidative stress, and angiogenesis in type 1 diabetic rat skin wound healing. J Nat Prod. 2013 Nov 22;76(11):2047-53. doi: 10.1021/np4002898. Epub 2013 Nov 7. PMID 24200239
- [Background] Dabrowski W, Gagos M, Siwicka-Gieroba D, Piechota M, Siwiec J, Bielacz M, Kotfis K, Stepulak A, Grzycka-Kowalczyk L, Jaroszynski A, Malbrain ML. Humulus lupus extract rich in xanthohumol improves the clinical course in critically ill COVID-19 patients. Biomed Pharmacother. 2023 Feb;158:114082. doi: 10.1016/j.biopha.2022.114082. Epub 2022 Dec 9. PMID 36508996
- [Background] Dartiguelongue JB. Systemic inflammation and sepsis. Part I: Storm formation. Arch Argent Pediatr. 2020 Dec;118(6):e527-e535. doi: 10.5546/aap.2020.eng.e527. English, Spanish. PMID 33231055
- [Background] Chong DLW, Sriskandan S. Pro-inflammatory mechanisms in sepsis. Contrib Microbiol. 2011;17:86-107. doi: 10.1159/000324022. Epub 2011 Jun 9. PMID 21659748
- [Background] Gaudette S, Smart L, Woodward AP, Sharp CR, Hughes D, Bailey SR, Dandrieux JRS, Santos L, Boller M. Biomarkers of endothelial activation and inflammation in dogs with organ dysfunction secondary to sepsis. Front Vet Sci. 2023 Jul 13;10:1127099. doi: 10.3389/fvets.2023.1127099. eCollection 2023. PMID 37520007
- [Background] Girisa S, Saikia Q, Bordoloi D, Banik K, Monisha J, Daimary UD, Verma E, Ahn KS, Kunnumakkara AB. Xanthohumol from Hop: Hope for cancer prevention and treatment. IUBMB Life. 2021 Aug;73(8):1016-1044. doi: 10.1002/iub.2522. Epub 2021 Jul 6. PMID 34170599
- [Background] Jung F, Staltner R, Tahir A, Baumann A, Burger K, Halilbasic E, Hellerbrand C, Bergheim I. Oral intake of xanthohumol attenuates lipoteichoic acid-induced inflammatory response in human PBMCs. Eur J Nutr. 2022 Dec;61(8):4155-4166. doi: 10.1007/s00394-022-02964-2. Epub 2022 Jul 20. PMID 35857130
- [Background] Lee IS, Lim J, Gal J, Kang JC, Kim HJ, Kang BY, Choi HJ. Anti-inflammatory activity of xanthohumol involves heme oxygenase-1 induction via NRF2-ARE signaling in microglial BV2 cells. Neurochem Int. 2011 Feb;58(2):153-60. doi: 10.1016/j.neuint.2010.11.008. Epub 2010 Nov 18. PMID 21093515
- [Background] Li F, Yao Y, Huang H, Hao H, Ying M. Xanthohumol attenuates cisplatin-induced nephrotoxicity through inhibiting NF-kappaB and activating Nrf2 signaling pathways. Int Immunopharmacol. 2018 Aug;61:277-282. doi: 10.1016/j.intimp.2018.05.017. Epub 2018 Jun 12. PMID 29906742
- [Background] Lin Y, Zang R, Ma Y, Wang Z, Li L, Ding S, Zhang R, Wei Z, Yang J, Wang X. Xanthohumol Is a Potent Pan-Inhibitor of Coronaviruses Targeting Main Protease. Int J Mol Sci. 2021 Nov 9;22(22):12134. doi: 10.3390/ijms222212134. PMID 34830015
- [Background] Luescher S, Urmann C, Butterweck V. Effect of Hops Derived Prenylated Phenols on TNF-alpha Induced Barrier Dysfunction in Intestinal Epithelial Cells. J Nat Prod. 2017 Apr 28;80(4):925-931. doi: 10.1021/acs.jnatprod.6b00869. Epub 2017 Feb 24. PMID 28234482
- [Background] Nolan A, Weiden MD, Thurston G, Gold JA. Vascular endothelial growth factor blockade reduces plasma cytokines in a murine model of polymicrobial sepsis. Inflammation. 2004 Oct;28(5):271-8. doi: 10.1007/s10753-004-6050-3. PMID 16134000
- [Background] Rahman SU, Ali T, Hao Q, He K, Li W, Ullah N, Zhang Z, Jiang Y, Li S. Xanthohumol Attenuates Lipopolysaccharide-Induced Depressive Like Behavior in Mice: Involvement of NF-kappaB/Nrf2 Signaling Pathways. Neurochem Res. 2021 Dec;46(12):3135-3148. doi: 10.1007/s11064-021-03396-w. Epub 2021 Aug 16. PMID 34398408
- [Background] Stevens JF, Page JE. Xanthohumol and related prenylflavonoids from hops and beer: to your good health! Phytochemistry. 2004 May;65(10):1317-30. doi: 10.1016/j.phytochem.2004.04.025. PMID 15231405
- [Background] Tang Z, Feng Y, Nie W, Li C. Xanthohumol attenuates renal ischemia/reperfusion injury by inhibiting ferroptosis. Exp Ther Med. 2023 Oct 24;26(6):571. doi: 10.3892/etm.2023.12269. eCollection 2023 Dec. PMID 37954118
- [Background] Xiao-Lei S, Tian-Shuang X, Yi-Ping J, Na-Ni W, Ling-Chuan X, Ting H, Hai-Liang X. Humulus lupulus L. extract and its active constituent xanthohumol attenuate oxidative stress and nerve injury induced by iron overload via activating AKT/GSK3beta and Nrf2/NQO1 pathways. J Nat Med. 2023 Jan;77(1):12-27. doi: 10.1007/s11418-022-01642-1. Epub 2022 Sep 8. PMID 36074228
- [Background] Xin G, Wei Z, Ji C, Zheng H, Gu J, Ma L, Huang W, Morris-Natschke SL, Yeh JL, Zhang R, Qin C, Wen L, Xing Z, Cao Y, Xia Q, Li K, Niu H, Lee KH, Huang W. Xanthohumol isolated from Humulus lupulus prevents thrombosis without increased bleeding risk by inhibiting platelet activation and mtDNA release. Free Radic Biol Med. 2017 Jul;108:247-257. doi: 10.1016/j.freeradbiomed.2017.02.018. Epub 2017 Feb 8. PMID 28188927
- [Background] Zhu L, Fan X, Cao C, Li K, Hou W, Ci X. Xanthohumol protect against acetaminophen-induced hepatotoxicity via Nrf2 activation through the AMPK/Akt/GSK3beta pathway. Biomed Pharmacother. 2023 Sep;165:115097. doi: 10.1016/j.biopha.2023.115097. Epub 2023 Jul 3. PMID 37406514